CLINICAL TRIAL: NCT06675422
Title: JY231 Injection for the Treatment of Active Systemic Lupus Erythematosus (SLE) - A Safety, Tolerability, and Efficacy Study
Brief Title: JY231 Injection for the Treatment of Active Systemic Lupus Erythematosus (SLE)
Acronym: JY231
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-24-005
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-09

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JY231 injection for the treatment of active systemic lupus erythematosus (Experimental)
  Interventions: Drug: JY231 injection

INTERVENTIONS:
Drug: JY231 injection — Dose escalation was carried out using the 3+3 principle and the mode of administration was intravenous.

SUMMARY:
Early exploratory clinical study of the safety, tolerability and initial efficacy of JY231 injection in the treatment of active systemic lupus erythematosus (SLE)

DETAILED DESCRIPTION:
This is a single-center, single-arm. open-label clinical study, in this study. approximately 10-20 patients with active systemic lupus erythematosus (SLE) will be enrolled for JY231 infusion therapy. The safety of JY231 was evaluated by observing adverse events after therapy. Evaluate the effectiveness of JY231 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with SLE according to the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria or the 2012 Systemic Lupus Erythematosus International Clinical Collaboration (SLICC) criteria.
2. Must have been treated with glucocorticoids in combination with immunosuppressants and/or biologics for at least 2 months prior to screening and have been dose stable for >2 weeks, with the disease remaining active (i.e., prior glucocorticoid + immunosuppressant or glucocorticoid + immunosuppressant + biologics, any of the above medications alone do not qualify). Oral corticosteroids must meet the following requirements: 1) Prednisone (or equivalent) ≥ 7.5 mg/day; 2) When used in combination with immunosuppressants and/or biologics, there is no minimum daily dose requirement for corticosteroids.
3. positive anti-nuclear antibody (ANA), and/or positive anti-ds-DNA antibody, and/or positive anti-Smith antibody at screening.
4. Screening Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score >6 and 'clinical' SLEDAI-2K score ≥4.

1)Note: 'Clinical' SLEDAI-2K is a SLEDAI-2K score that excludes scores attributable to any urine or laboratory findings, including immunological indicators: 2)-Includes scores for the following clinical items: arthritis, myositis, rash, alopecia, mucosal ulcers, pleurisy, pericarditis, or vasculitis; 3)-excludes scores attributable to fever, SLE headache and organic brain syndromes.

5.British Isles Lupus Assessment Group 2004 (BILAG2004) score of at least one of the following:

1. ≥1 organ system BILAG2004 grade A disease
2. ≥2 organ system BILAG2004 Grade B disorders 6.Physician's General Assessment (PGA) score of ≥1.0 (0-3 visual analogue scale VAS) at screening.

Exclusion Criteria:

1. Combination of other autoimmune diseases requiring systemic therapy.
2. SLE patients: the presence of still uncontrolled lupus crisis within 8 weeks prior to screening, including acute progressive lupus nephritis, severe neuropsychiatric lupus, severe haemolytic anaemia, severe immune thrombocytopenia, granulocyte deficiency, severe cardiac damage, severe lupus pneumonitis, severe lupus hepatitis, severe vasculitis, etc., which were assessed as unsuitable for participation in the study by the investigator.
3. Pre-screening comorbidity with clinically significant central nervous system disease or pathological changes not due to lupus, including but not limited to: cerebral vascular accident, aneurysm, epilepsy, convulsions/convulsions, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndromes, or psychosis.
4. History of allogeneic bone marrow or stem cell transplantation or solid organ transplantation (e.g., kidney, lung, heart, liver) or future plans for such transplantation.
5. Presence of clinically significant cardiovascular dysfunction in the 12 months prior to screening, including, but not limited to: class III or IV heart failure as defined by the New York Heart Association (NYHA), myocardial infarction, unstable angina pectoris, uncontrolled or symptomatic atrial arrhythmia, any ventricular arrhythmia.
6. Presence of significant pulmonary or cardiac manifestations such as pericarditis, pleural effusion at the time of screening, assessed by the investigator to be unsuitable for participation in this study.
7. Patients with severe asthma or chronic obstructive pulmonary disease (COPD), mild or moderate asthma or COPD on stable therapy may be enrolled.
8. History of malignancy within 5 years prior to signing the Informed Consent Form (ICF), except adequately treated or surgically resected, non-melanoma skin cancers or carcinoma in situ (e.g., cervical cancer, bladder cancer, breast cancer) without residual disease.
9. Women who are pregnant or breastfeeding.
10. History of recurrent infections requiring hospitalisation and intravenous antibiotics (e.g. 3 or more episodes of the same type of infection in the past 1 year).
11. Active infection requiring systemic treatment, such as infectious pneumonia, tuberculosis, etc., within 2 weeks prior to clearance.
12. Hepatitis B surface antigen (HBsAg) positive, or Hepatitis B core antibody (HBcAb) positive and peripheral blood Hepatitis B Virus (HBV) DNA test positive; Hepatitis C Virus (HCV) antibody positive and peripheral blood HCV RNA positive; human immunodeficiency virus (HIV) antibody positive; syphilis antibody positive.
13. Have received a live attenuated vaccine within 4 weeks prior to clearance or plan to receive a live attenuated vaccine during the course of the study.
14. Have received high-dose corticosteroids (prednisone ≥ 60 mg/day or equivalent) within 4 weeks prior to clearance, or are unable to taper prednisone to ≤ 10 mg/day 5 days prior to clearance.
15. Inability to taper or elute background therapy prior to clearing chemotherapy as described in Table 3.
16. Receiving renal replacement therapy within 3 months prior to screening or anticipating the need for renal replacement therapy during the study.
17. History of drug or alcohol abuse within 1 year prior to screening.
18. History or evidence of suicidal thoughts within 6 months prior to screening or any suicidal behaviour within the previous 12 months that the investigator considers to be a significant risk of suicide.
19. Use of another study drug within 4 weeks or 5 half-lives (whichever is longer) prior to screening.
20. History of hypersensitivity or life-threatening reaction to the study drug or any component or preparation of the study treatment (including clear chemotherapy). See the Investigator's Brochure (IB) for more information about the components of the study drug.
21. Any condition that, in the opinion of the investigator, may affect participation in the study, pose a safety risk to patients, or may confound the interpretation of study results.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From enrollment to the end of treatment at 6 months

SECONDARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | Up to 12 months after infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Doctor, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th HJointLogistics, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No